CLINICAL TRIAL: NCT01630148
Title: Bemiparin as a Thromboprophylaxis After Benign Gynaecological Surgeries:A Randomized Clinical Trial
Brief Title: Bemiparin as a Thromboprophylaxis After Gynaecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, SHAHLA KAREEM ALALAF, Assistant Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMU
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Deep Vein Thrombosis (DVT); Pulmonary Embolism
Keywords: Thromboprophylaxis; Bemiparin; Low Molecular Weight Heparin; Major Gynaecological Surgeries; Benign Gynaecological Surgeries
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — bemiparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bemiparin (Active Comparator): group one will be women who are risky for venous thromboembolic diseases after benign gynaecological surgeries, each will receive Bemiparin
  Interventions: Drug: Bemiparin
- control group (No Intervention): women will undergo benign gynaecological surgeries and are risky for venous thrombosis, they will not receive any intervention. The patients will be followed up to 30 days after surgery.

INTERVENTIONS:
Drug: Bemiparin — Bemiparin Sodium 3,500IU anti Xa/0.3 ml solution for injection in pre-filled syringe will be provided for each patient in Bemiparin group (Moderate, High and Highest risk groups for thromboembolism) 6 hours after surgery and then daily for up to 7 days.
  Other Names: Hibor; Laboratories Rovi pharmaceuticals
  Arms: Bemiparin

SUMMARY:
The use of prophylaxis for venous thromboembolism (VTE) remains grossly underused for women who undergo gynecologic surgery for benign conditions world wide and especially in developing countries including our region. Having a research in our locality for the first time might raise awareness of the importance of VTE prophylaxis.

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) and pulmonary embolism (PE), also referred to as venous thromboembolic events (VTE), are two major complications after gynaecological surgeries that can result in significant morbidity and mortality. The incidence of VTE after gynaecologic surgery varies depending on the method used for diagnosis. The rate of clinical DVT is estimated to be 3% after gynaecological surgery if no thromboprophylaxis was used. The rate of VTE assumed to decrease to 0.4% if Low molecular weight heparin was used as a thromboprophylaxis.

According to our knowledge there are no published researches on the effect of the new second generation Low molecular Weight Heparin Bemiparin as a thromboprophylaxis after benign gynaecological surgery in comparison to a control group.

ELIGIBILITY:
Inclusion Criteria:

* female undergoing Benign gynecological surgeries.
* Having moderate,high and very high risk factors for venous thromboembolism.
* No contraindications for the use of Heparin.

Exclusion Criteria:

* Having mild risk factors for thromboembolism.
* Active vaginal bleeding.
* Thrombocytopaenia.
* any patient who is already on anticoagulant.
* Sever renal or Liver diseases.

Ages: 15 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evidences of clinical thromboembolic disease after gynaecological surgeries | within the first 30 days after surgery the first 30 days
  to determine the efficacy of the new second generation LMWH in prevention Deep vein thrombosis and pulmonary embolism after gynaecological surgeries

SECONDARY OUTCOMES:
to determine the side effects of Bemiparin injection | after receiving the injections and up to 30 days after surgery
  To determine the safety of Bemiparin after gynaecological surgeries including bruising or pain at site of injection,itching,allergic skin reactions,urticaria, bleeding,

CONTACTS AND LOCATIONS:
Overall Officials: Shahla K. Alalaf, M.D, Principal Investigator — Hawler Medical University; Ariana K. Jawad, C.A.B.OG, Study Chair — Hawler Ministry of Health; Rojan K. Jawad, Diploma, Study Chair — Hawler Medical University; Mahabad S. Ali, Diploma, Study Chair — Hawler Ministry of Health; Namir G. Al Tawil, Professor, Study Director — Hawler Medical University
Locations (1):
- Shahla Kareem Alalaf, Erbil, Kurdistan Region, Iraq